CLINICAL TRIAL: NCT05969834
Title: Human Chorionic Gonadotropin Levels After Ovulation Triggering as Predictors of Intracytoplasmic Sperm Injection Outcome
Brief Title: HCG Levels After Ovulation Triggering as Predictors of ICSI Outcome
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: MD.20.09.370
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Infertility
Keywords: Ovulation triggering; uHCG; rHCG; GnRH; Dual trigger
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin; Triptorelin Pamoate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- uHCG group: Trigger intramuscular (IM) administration of 10000 IU of uHCG
  Interventions: Drug: uHCG
- rHCG group: Trigger with subcutaneous (SC) administration of 6500 IU of rHCG
  Interventions: Drug: rHCG
- Dual trigger group: Combined SC administration of 0.1 mg of GnRHa and IM administration of 2500 IU of uHCG
  Interventions: Drug: uHCG and GnRHa

INTERVENTIONS:
Drug: uHCG — Final oocyte maturation will be triggered by IM administration of 10000 IU of uHCG (Choriomon)
  Other Names: Choriomon
  Groups: uHCG group
Drug: rHCG — Final oocyte maturation will be triggered by SC administration of 6500 IU of rHCG (Ovitrelle)
  Other Names: Ovitrelle
  Groups: rHCG group
Drug: uHCG and GnRHa — Final oocyte maturation will be triggered by combined SC administration of 0.1 mg of GnRHa (Decapeptyl, Triptorelin) and IM administration of 2500 IU of uHCG (Choriomon)
  Other Names: Decapeptyl and Choriomon
  Groups: Dual trigger group

SUMMARY:
This study aimed to assess the correlation between HCG levels after ovulation triggering and ICSI outcomes, affected by HCG formulation and dose

DETAILED DESCRIPTION:
The aims of this study are:

1. To assess the correlation between serum human chorionic gonadotropin (hCG) level after ovulation triggering and intracytoplasmic sperm injection (ICSI) outcome including: oocyte maturity and quality, good quality embryo rate, blastocyst formation rate and pregnancy rate
2. To determine if there is an association between type and dose of the trigger and ICSI outcome.

ELIGIBILITY:
Inclusion Criteria:

* Women who will undergo controlled ovarian stimulation (COS) through fixed GnRH antagonist protocol

Exclusion Criteria:

* BMI > 30 kg/m2
* Irregular menstruation
* Severe male factor abnormality
* Poor ovarian reserve
* Endometriosis
* Uterine abnormality

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who will undergo controlled ovarian stimulation (COS) through fixed GnRH antagonist protocol with ovulation triggering, according to the risk of OHSS, by: 1) urinary HCG (uHCG); 2) recombinant HCG (rHCG); or 3) a combination of GnRHa and HCG (dual trigger)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-08-07 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6 weeks after embryo transfer
  Number of clinical pregnancies (defined as presence of at least one intrauterine gestational sac with fetal pole and cardiac activity on TVS scan at 4-6 weeks after the ET) divided by the number of ET procedures

SECONDARY OUTCOMES:
Oocyte maturation rate | On 1 day of oocyte retrieval
  Number of mature oocytes divided by the number of retrieved oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Engy Abdallah, MSc, Principal Investigator — Mansoura University; Mohamed S Abdelhafez, MD, Study Director — Mansoura University; Mohamed Elzayat, MD, Study Chair — Royal Center; Amoura Abou-ElNaga, MD, Study Chair — Mansoura University
Locations (1):
- Royal Center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided